CLINICAL TRIAL: NCT01244308
Title: Effectiveness and Reliability of VectSelect™ Feature for Avoidance of Phrenic Nerve Stimulation in CRT Patients
Brief Title: Effectiveness and Reliability of VectSelect™ Feature for Avoidance of Phrenic Nerve Stimulation in Cardiac Resynchronisation Therapy (CRT) Patients
Acronym: Efface
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: T86
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Phrenic nerve stimulation; LV pacing configuration; CRT; Cardiac resynchronisation therapy; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It's the aim of this study to analyse efficacy and reliability of VectSelect Feature for avoidance of phrenic nerve stimulation in cardiac resynchronisation therapy (CRT) patients.

ELIGIBILITY:
Inclusion Criteria:

* indication for CRT-D implantation / upgrade
* written informed consent

Exclusion Criteria:

* pregnancy
* age < 18 years
* patients, who cannot visit the routine follow ups (within first 3.5months)
* participants to other studies with active treatment arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for implantation of CRT-D device
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Amount of patients with at least one acceptable LV pacing configuration. | First Follow Up after hospital discharge (approx. 1-3 months)
  Amount of patients with at least one acceptable, programmable LV pacing configuration. Definition of acceptable LV pacing configuration: LV pacing threshold <=2.5V@0.5ms AND Phrenic nerve threshold is at least twice as high as LV pacing threshold AND LV pacing impedance >=200 Ohms.
  Only patients with implanted CRT-D and bipolar leftventricular lead are taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Klein, Dr. med., Principal Investigator — Universitätsklinikum Leipzig AÖR
Locations (10):
- Germany (10):
  - Medizinische Einrichtungen der RWTH Aachen, Aachen
  - Hufeland Klinikum GmbH, Bad Langensalza
  - Cardioangiologisches Centrum Bethanien, Frankfurt am Main
  - Universitätsklinikum Gießen und Marburg GmbH Sitz Gießen, Giessen
  - Universitäres Herzzentrum Hamburg GmbH (UHZ), Hamburg
  - Katholisches Krankenhaus Marienhospital Universitätsklinik, Herne
  - Klinikum Kassel gGmbH, Kassel
  - Universitätsklinikum Leipzig AÖR, Leipzig
  - Niels-Stensen-Kliniken Marienhospital, Osnabrück
  - Klinikum Dorothea Christiane Erxleben GmbH, Quedlinburg

REFERENCES:
- [Result] Klein N, Klein M, Weglage H, Przibille O, Fischer S, Trappe HJ, Birkenhauer F, Pfeiffer D; Efface Phrenic Stim Study Group. Clinical efficacy of left ventricular pacing vector programmability in cardiac resynchronization therapy defibrillator patients for management of phrenic nerve stimulation and/or elevated left ventricular pacing thresholds: insights from the Efface Phrenic Stim study. Europace. 2012 Jun;14(6):826-32. doi: 10.1093/europace/eur412. Epub 2012 Jan 25. PMID 22277645